CLINICAL TRIAL: NCT04844164
Title: Prospective Non-randomised Controlled Study of Vitamin D Metabolism in Patients With Endocrine Disorders (Acromegaly, Cushing's Disease, Primary Hyperparathyroidism, Diabetes Mellitus Type 1) Treated With Cholecalciferol Bolus Dose
Brief Title: Vitamin D Metabolism in Patients With Endocrine Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocrinology Research Centre, Moscow (Other Government)
Collaborators: Russian Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ERC_2021/01; 19-15-00243 (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Pituitary ACTH Hypersecretion; Acromegaly; Diabetes Mellitus, Type 1; Primary Hyperparathyroidism
Keywords: Vitamin D; Vitamin D deficiency; Chromatography, Liquid; Tandem Mass Spectrometry; Cholecalciferol
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Acromegaly; Diabetes Mellitus, Type 1; Hyperparathyroidism, Primary; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cushing's Disease (Experimental)
  Interventions: Drug: Cholecalciferol 15000 UNT/ML Oral Solution
- Acromegaly (Experimental)
  Interventions: Drug: Cholecalciferol 15000 UNT/ML Oral Solution
- Diabetes Mellitus Type 1 (Experimental)
  Interventions: Drug: Cholecalciferol 15000 UNT/ML Oral Solution
- Primary Hyperparathyroidism (Experimental)
  Interventions: Drug: Cholecalciferol 15000 UNT/ML Oral Solution
- Control group (Experimental)
  Interventions: Drug: Cholecalciferol 15000 UNT/ML Oral Solution

INTERVENTIONS:
Drug: Cholecalciferol 15000 UNT/ML Oral Solution — A single dose (150,000 IU) of cholecalciferol aqueous solution per os

SUMMARY:
This prospective controlled interventional study aims to reveal the diversity of vitamin D metabolism in patients with certain endocrine disorders (Cushing's disease, acromegaly, primary hyperparathyroidism, diabetes mellitus type 1) compared to healthy adults. All patients will receive a single dose (150,000 IU) of cholecalciferol aqueous solution orally. Laboratory assessments including serum vitamin D metabolites (25(OH)D3, 25(OH)D2, 1,25(OH)2D3, 3-epi-25(OH)D3, 24,25(OH)2D3 and D3), free 25(OH)D, vitamin D-binding protein (DBP) and parathyroid hormone (PTH) as well as serum and urine biochemical parameters will be performed before the intake and on Days 1, 3 and 7 after the administration.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis (arms "Cushing's Disease", "Acromegaly", "Diabetes Mellitus Type 1", "Primary Hyperparathyroidism")
* active phase of the disease (arms "Cushing's Disease", "Acromegaly")
* no history of surgical and specific pharmacological treatment (arm "Primary Hyperparathyroidism")
* HbA1c <8.0% (arm "Diabetes Mellitus Type 1")
* absence of the specified endocrine disorders (arm "Control group")

Exclusion Criteria:

* factors associated with vitamin D level

  * intake of the following drugs during the 3 months preceding the study: vitamin D medications; glucocorticosteroids; antiretroviral drugs; antifungal drugs; cholestyramine, orlistat; antiepileptic drugs; antidepressants (fluoxetine); diuretics (spironolactone); antimicrobial agents (macrolides, tetracyclines, isoniazid, rifampin, primaquine); chemotherapy (cyclophosphamide, tamoxifen, paclitaxel, ifosfamide, irinotecan, etoposide, vinblastine); immunosuppressants (cyclosporin A, tacrolimus, sirolimus); H2 receptor antagonists.
  * BMI >35 kg/m2
  * pregnancy
  * granulomatous disease (sarcoidosis, tuberculosis, histoplasmosis, berylliosis, coccidiomycosis)
  * disease with malabsorption syndrome (Crohn's disease, ulcerative colitis, celiac disease, post-bariatric surgery condition, decompensation of chronic pancreatitis)
  * reduced renal function (eGFR <60 ml/min/1.73m2)
  * laboratory signs of liver failure (hypoalbuminemia, hypoprothrombinemia)
* hypercalcemia or risk factors for hypercalcemia

  * serum total calcium >3.0 mmol/L
  * myeloma
  * immobilization
  * thiazide diuretics intake
* allergy to vitamin D drugs
* total 25(ОН)D >60 ng/ml (determined by chemiluminescent immunoanalysis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 261 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Baseline 25(OH)D3 level | Day 0
  Measured in ng\mL.
Change in 25(OH)D3 level | Day 1, 3, 7
  Measured in ng\mL.

SECONDARY OUTCOMES:
Serum total calcium | Day 0, 1, 3, 7
  Measured in mmol\L
Serum albumin-adjusted calcium | Day 0, 1, 3, 7
  Measured in mmol\L
Serum phosphorus | Day 0, 1, 3, 7
  Measured in mmol\L
Serum PTH | Day 0, 1, 3, 7
  Measured in pg/mL
Serum creatinine | Day 0, 1, 3, 7
  Measured in μmol/L
Serum albumin | Day 0, 1, 3, 7
  Measured in g/L
Serum magnesium | Day 0, 1, 3, 7
  Measured in mmol\L
Calcium-creatinine ratio in spot urine | Day 0, 1, 3, 7
  Measured in mmol/mmol
Phosphorus-creatinine ratio in spot urine | Day 0, 1, 3, 7
  Measured in mmol/mmol
1,25(OH)2D3 level | Day 0, 1, 3, 7
  Measured in pg\mL.
24,25(OH)2D3 level | Day 0, 1, 3, 7
  Measured in ng\mL.
3-epi-25(OH)D3 level | Day 0, 1, 3, 7
  Measured in ng\mL.
25(OH)D2 level | Day 0, 1, 3, 7
  Measured in ng\mL.
D3 level | Day 0, 1, 3, 7
  Measured in ng\mL.
25(OH)D3/24,25(OH)2D3 ratio | Day 0, 1, 3, 7
25(OH)D3/1,25(OH)2D3 ratio | Day 0, 1, 3, 7
Serum free 25(OH)D | Day 0, 1, 3, 7
  Measured in pg/mL
Serum vitamin D-binding protein | Day 0, 1, 3, 7
  Measured in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Liudmila Rozhinskaya, MD, PhD, Principal Investigator — Endocrinology Research Centre, Moscow
Locations (1):
- Endocrinology Research Centre, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Povaliaeva A, Pigarova E, Zhukov A, Bogdanov V, Dzeranova L, Mel'nikova O, Pekareva E, Malysheva N, Ioutsi V, Nikankina L, Rozhinskaya L. Evaluation of Vitamin D Metabolism in Patients with Type 1 Diabetes Mellitus in the Setting of Cholecalciferol Treatment. Nutrients. 2020 Dec 18;12(12):3873. doi: 10.3390/nu12123873. PMID 33352890
- [Derived] Povaliaeva AA, Bogdanov VP, Zhukov AY, Pigarova EA, Dzeranova LK, Rozhinskaya LY, Mel'nichenko GA, Mokrysheva NG. Characterization of vitamin D metabolism in active acromegaly in the setting of bolus (150,000 IU) cholecalciferol treatment. Endocrine. 2022 May;76(2):407-418. doi: 10.1007/s12020-022-02994-0. Epub 2022 Feb 9. PMID 35138562